CLINICAL TRIAL: NCT04041999
Title: Randomized Study of a Daily Cognition Training Program Versus Traditional Cognitive Stimulation in Older Adults
Brief Title: Study of a Daily Cognition Training Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, Prof. Dr. Eduardo J Fernández Rodríguez, PhD. Occupational therapy. University of Salamanca., University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 000263
Record Dates: First submitted 2019-07-22; First posted 2019-08-01 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Occupational Therapy; Cognition Disorders in Old Age; Cognitive Dysfunction; Rehabilitation
Keywords: Occupational therapy; cognition; rehabilitation
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Experimental, randomized, stratified, prospective, longitudinal study using a parallel scheme of fixed allocation experimental group and control group
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Daily Cognition Training Program (Experimental): The intervention was administered by a qualified professional, in this case an occupational therapist. And it was always individually through specific activities or exercises.
  Tasks are carried out in which the subject has to exercise different cognitive functions (praxies, attention, language, memory orientation, gnosias and executive functions; mainly working memory decision making, planning, reasoning and temporal estimation) during the development of AIVD For this, similar materials are used to those that the elderly could find in daily tasks or when solving day-to-day problems.
  Specifically we focus on tasks related to taking medication and adherence to treatment.
  Interventions: Behavioral: Daily Cognition Training Program
- Traditional Cognitive Stimulation Program (Active Comparator): The intervention was administered by a qualified professional, in this case an occupational therapist. And it was always individually through specific activities or exercises.
  Tasks are performed to work various cognitive functions.
  Interventions: Behavioral: Daily Cognition Training Program

INTERVENTIONS:
Behavioral: Daily Cognition Training Program — Tasks are carried out in which the subject has to exercise different cognitive functions (praxies, attention, language, memory orientation, gnosias and executive functions; mainly working memory decision making, planning, reasoning and temporal estimation) during the development of AIVD For this, similar materials are used to those that the elderly could find in daily tasks or when solving day-to-day problems.
  Specifically we focus on tasks related to taking medication and adherence to treatment. Some examples of tasks are: the management of a medical prescription, expiration of a medication, understanding of the prescriptions made by the doctor, guidelines for taking medication (doses, schedules ...) and indications and contraindications, filling pill boxes, recall of controls doctors, medication control, prospective memory of medical management, etc.

SUMMARY:
HYPOTHESIS In older adults who receive a direct intervention from the perspective of occupational therapy with a "Training Program in Daily Cognition", there are greater benefits, both in the overall cognitive performance and in the levels of daily cognition, that in the older adults who receive an intervention based on a "Traditional Cognitive Stimulation Program", achieving not only an improvement or maintenance of cognitive functions, but a generalization and transfer of that improvement in their daily lives and occupational performance.

OBJECTIVES: To evaluate the effectiveness of a "Training Program in Daily Cognition" in the elderly, to improve the levels of daily cognition and global cognitive performance.

SPECIFIC OBJECTIVES:

Compare the difference in levels of daily cognition between the participants of the control group who carry out a "Traditional Cognitive Stimulation Program" and the participants of the experimental group who carry out a "Training Program in Daily Cognition".

Analyze if there is a difference in the levels of global cognitive performance between the participants of the control group that carry out a "Traditional Cognitive Stimulation Program" and the participants of the experimental group that carry out a "Training Program in Daily Cognition".

To study the relationship between standard psychometric tests that measure cognitive performance and the ECB Daily Cognition Battery Recognition Test that measures daily cognition.

Analyze if there is a relationship between age and cognitive performance and the daily cognition of the elderly.

Describe the relationship between the educational level that the participants possess and the cognitive performance and their daily cognition Evaluate the impact of gender in the elderly with cognitive performance and daily cognition.

Check whether or not physical activity influences the cognitive performance and daily cognition of study participants.

STUDY DESIGN: Experimental, randomized, stratified, prospective, longitudinal study using a parallel scheme of fixed allocation experimental group and control group.

The protocol has been authorized by the Ethics Committee of the Salamanca health area to make the project possible.

DETAILED DESCRIPTION:
OBJECTIVES To evaluate the effectiveness of a "Training Program in Daily Cognition" in the elderly, to improve levels of daily cognition and overall cognitive performance.

SPECIFIC OBJECTIVES:

* Compare the difference in levels of daily cognition between the participants of the control group who carry out a "Traditional Cognitive Stimulation Program" and the participants of the experimental group who carry out a "Training Program in Daily Cognition".
* To analyze if there is a difference in the levels of global cognitive performance between the participants of the control group that carry out a "Traditional Cognitive Stimulation Program" and the participants of the experimental group that carry out a "Training Program in Daily Cognition".
* To study the relationship between the standard psychometric tests that measure cognitive performance and the Recognition Test (Declarative Memory) of the ECB Daily Battery of Cognition (Everday Cognition Battery), which measures daily cognition.
* Analyze if there is a relationship between age and cognitive performance and the daily cognition of the elderly.
* Describe the relationship between the educational level of the participants and cognitive performance and their daily cognition
* Evaluate the impact of gender on the elderly with performance Cognitive and everyday cognition.
* Check whether or not physical activity influences cognitive performance and daily cognition of study participants.

STUDY DESIGN Experimental, randomized, stratified, prospective, longitudinal study using a parallel scheme of fixed allocation experimental group and control group; in which the evolution of cognitive performance in individuals who voluntarily enrolled in the Occupational Therapy Program offered by HE. Salamanca City Council in different Senior Centers in the city of Salamanca.

The study was carried out over four years with three phases without intervention between them. Each intervention phase lasted 12 weeks. Participants were assessed at the beginning and at the end of each intervention period.

The realization of this research study in older adults was approved by the Bioethics Committee of the University of Salamanca.

SITE

The scope of the study was ten Senior Centers belonging to HE. Salamanca City Council, participating in the Occupational Therapy Program, which is carried out by the Department of Physiotherapy of the University of Salamanca.

SAMPLE SELECTION Population under study The study involved healthy older adults, of both sexes, not institutionalized, from the town of Salamanca who voluntarily carried out the Occupational Therapy Program, taught from the University of Salamanca, in its corresponding Senior Center, during the years 2014- 2018.

RANDOMIZATION The randomization process of the groups of participants was carried out with respect to the order of the centers where the program was carried out. It was carried out by the simple random assignment method, for this a random number table generated using the Microsoft Excel 2016R program was used. By means of said random number table, the centers that obtain an even number from the experimental group were assigned to the centers that obtained an odd number from the control group.

SAMPLE SIZE The sample of the study was formed by all users of the different centers of greater affiliation to the Occupational Therapy Program offered from the University of Salamanca, who met the inclusion / exclusion criteria, who authorized their participation in the study voluntarily, through the signature of an informed consent.

INDEPENDENT VARIABLES:

- Direct intervention from the perspective of occupational therapy in the improvement of daily cognition through a "Daily Cognition Training Program".

DEPENDENT VARIABLES:

* Daily cognition: Measured with the Everyday Cognition Battery (ECB).
* Cognitive performance: Measured with the Rapid Evaluation of Cognitive Functions (ERFC). The ERFC in addition to a total score will provide us with other variables that are: Temprospatial orientation, attention and memory, mental calculation, reasoning and judgment, similarities, comprehension, denomination, repetition, written order, verbal fluency, praxies, visual recognition and writing.

INTERVENING VARIABLES:

* Age
* sex
* Level of studies
* Physical activity DATA ASSESSMENT AND COLLECTION INSTRUMENTS As indicated in detail later in the process description section, each participant carried out a total of 8 assessments, 2 for each of the 4 of the intervention phases. An initial and another final. The first assessment of the study coincides with the assessment of the beginning of the Occupational Therapy Program for the 2014-2015 period, and the last assessment corresponds to the assessment of the end of the 2017-2018 program. The evaluations were carried out by five qualified occupational therapists, of which only one subsequently performed the intervention. In this way it is achieved that 80% of the evaluations are carried out by an external evaluator, to control, as far as possible, possible interferences or biases in the results.

To evaluate the different types of variables, the following registration sheets, scales and questionnaires have been used.

DEPENDENT VARIABLES:

For the dependent variables, in both groups, participants will be evaluated with two heteroadministered questionnaires; the Everyday Cognition Battery (ECB) Test and the Rapid Assessment of Cognitive Functions (ERFC) Test.

DESCRIPTION OF THE INTERVENTION Process description

1. First, participants interested in carrying out the Occupational Therapy Program must submit an access request, voluntarily registering in the corresponding Senior Center.

   In the period from May to June, the Department of Elders of the City of Salamanca proceeds to collect these requests from the elderly, from the Associations of Elders of the municipality who wish to participate in the following course in the Occupational Therapy Program. In the Municipal Centers for the Elderly "Juan de la Fuente" and "Tierra Charra" the call for applications is held approximately one month before the program begins.
2. After acceptance of admission to the program, the sample is determined taking into account that participants of the Occupational Therapy Program meet the inclusion and exclusion criteria previously established to participate in the study.
3. Delivery and reading of the participant information sheet (ANNEX 4), where all the questions about the study and the tests and scales that will be carried out in the assessments are explained. After the clarifications requested, the informed consent is read and signed (ANNEX 5) if they agree to be part of the study.
4. Assignment of groups randomly belonging to the experimental group or the control group.
5. Initial Assessment or Assessment 1 (V-1): performed before beginning the intervention by qualified occupational therapists. This assessment is the same both in the experimental group and in the control group and consists in formalizing the clinical history and in carrying out the tests indicated above that assess the cognitive performance of the participants.
6. Intervention phase 1 (FI-1): with a total of 20 sessions, making 2 weekly sessions, which is approximately 3 months long. Being annually the work period from October to May. Taking into account that it is intervened in 10 groups: In total, 200 work sessions are held distributed in 20 sessions in each of the 10 groups. FIGURE 6 shows the distribution over time of the different groups. 7) At the end of this intervention period, Valuation 2 (V-2) is carried out, consisting of the same tests that are performed on V-1. The time between V-1 and V-2 is the 1st STAGE.

8) After V - 2, in each center, a period is established in which participants do not receive intervention. We will call this period Phase of non-intervention 1 (FNI-1).

Each period of non-intervention lasts approximately one year. And in each center (FIGURE 7).

9) The 2nd STAGE begins with Assessment 3 (V-3), followed by Intervention Phase 2 (FI-2), and ends with Assessment 4 (V-4).

10) The process continues with the Non-intervention Phase 2 (FNI-2), which gives way to the 3rd STAGE; which begins with Assessment 5 (V-5), continues with intervention phase 3 (FI-3) and ends with Assessment 6 (V-6).

11) We would continue with the Non-intervention Phase 3 (FNI-3), reaching the last stage of the study, 4th STAGE. This stage is comprised of Assessment 7 (V-7), an Intervention Phase 4 (FI-4), and the last evaluation, which is Assessment 8 or Final Assessment (V-8).

In the 10 intervention groups the same scheme is followed. Each of the four intervention phases has an identical duration of approximately 3 months with 20 sessions. The three phases of non-intervention are 1 year each.

Description of the intervention The intervention is carried out in 10 groups, with the timing that we have seen previously.

In each group there are 2 sessions per week on random days, with a duration of 60 minutes, each group receiving a total of 20 sessions. In total, 200 intervention sessions are distributed in 20 sessions in each of the 10 groups, in each intervention phase. As in total, 4 intervention phases are carried out in the study: 800 intervention sessions are carried out.

The intervention sessions differ in terms of the procedures used in the experimental group and the control group.

A. Control group: An intervention is carried out based on a "Traditional Cognitive Stimulation Program".

· In the "Traditional Cognitive Stimulation Program", tasks are carried out to work various cognitive functions: orientation, gnosias, executive functions (mainly working memory decision making, planning, reasoning and temporal estimation), praxies, attention, language and memory .

B. Experimental group: An intervention is carried out based on a "Daily Cognition Training Program". Tasks are carried out in which the subject has to exercise different cognitive functions (praxies, attention, language, memory orientation, gnosias and executive functions; mainly working memory decision making, planning, reasoning and temporal estimation) during the development of AIVD For this, similar materials are used to those that the elderly could find in daily tasks or when solving day-to-day problems.

ETHICAL-LEGAL ASPECTS OF THE PROJECT The protocol has been authorized by the Ethics Committee of the Salamanca health area to make the project possible.

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 60 years of age and voluntarily enroll in the Occupational Therapy Program.
2. Be accepted in the Occupational Therapy Program.
3. Perform the initial assessment.
4. Voluntarily authorize their participation in the study, by signing an informed consent.

Exclusion Criteria:

1. Present cognitive impairment with clinical diagnosis.
2. Not have numerical and literacy skills.
3. Do not authorize your participation in the study.
4. Participate in some other cognitive stimulation program regularly.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Cognitive function | Up to 3 years
  Rapid evaluation of cognitive functions (ERFC)
Everyday cognition | Up to 3 years
  Everyday Cognition Battery (ECB)

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo José Fernández Rodríguez, PhD, Principal Investigator — University of Salamanca
Locations (1):
- Eduardo José Fernández Rodríguez, Salamanca, España, Spain

IPD SHARING:
Plan to Share IPD: Yes
A specific database will be created to which any external researcher can access after contact by email to the email edujfr@usal.es
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: We do not establish a specific period of time, access will be permanent.
Access Criteria: Investigador previa invitación por correo

REFERENCES:
- [Derived] Gomez CS, Rodriguez EJF. The effectiveness of a training programme in everyday cognition in healthy older adults: a randomised controlled trial. BMC Geriatr. 2021 Jan 28;21(1):79. doi: 10.1186/s12877-020-01998-7. PMID 33509113